CLINICAL TRIAL: NCT05076721
Title: The Role of Simulation-Based Training to Improve Team Performance in Implementing One Sepsis Hour Bundle in Intensive Care Unit
Brief Title: Effectiveness of Simulation Based Training in Implementing One Hour Bundle Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Adhrie Sugiarto, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IndonesiaUAnes117
Record Dates: First submitted 2021-09-18; First posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-09

CONDITIONS: Medical Education; Simulation Training; Sepsis
Keywords: medical education; simulation training; sepsis; high-fidelity manikin; one-hour bundle sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simulation group (Experimental): The simulation training group will receive a simulation training of a sepsis case which will see the participants implementing one-hour bundle sepsis with a high-fidelity manikin.
  Interventions: Other: Simulation training
- Conventional group (Experimental): The conventional training group will receive a case-based discussion of a sepsis case which will see the participants implementing one-hour bundle sepsis.
  Interventions: Other: Case-based discussion training

INTERVENTIONS:
Other: Simulation training — The participants in the simulation group will receive simulation training with high-fidelity manikin to practice and implement one-hour bundle sepsis
  Arms: Simulation group
Other: Case-based discussion training — The participants in the conventional group will only do a case-based discussion in implementing one-hour bundle sepsis
  Arms: Conventional group

SUMMARY:
This study aimed to compare simulation training with conventional training (case-based discussion only) to improve team performance in implementing one-hour sepsis bundle in the intensive care unit

DETAILED DESCRIPTION:
This was an experimental randomized single-blind study to examine the role of simulation-based training in improving team performance in conducting sepsis management. Subjects were sixteen doctors and twenty-four nurses working in the intensive care unit. The subjects were randomly divided into two treatment groups: the discussion group and the simulation group. Each treatment group was further divided into four small groups consisting of two doctors and three nurses. Prior to the training, every subject received a pretest for cognitive evaluation and a posttest at the end of the training. The performance of both groups in implementing one-hour sepsis bundle was assessed by solving a sepsis case in high fidelity manikin.

ELIGIBILITY:
Inclusion Criteria:

* Doctors working in Dr. Cipto Mangunkusumo Public Hospital's ICU
* Nurses working in Dr. Cipto Mangunkusumo Public Hospital's ICU

Exclusion Criteria:

* Doctors and nurses who are not fit or healthy to undergo this training

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-08-22 (Actual); Primary Completion 2020-10-24 (Actual); Study Completion 2020-10-24 (Actual)

PRIMARY OUTCOMES:
Differences in score of skills in implementing one-hour bundle sepsis in the intensive care unit assessed with checklist which were designed by four anesthesiologist-intensivists | upon study completion, in 1 day
  Measured by checklist which were designed by four anesthesiologist-intensivists before the study was conducted and validated by Aiken coefficient. The Aiken coefficient for this checklist were all >0.3 which is declared valid.

SECONDARY OUTCOMES:
Differences in intrateam communication's score in implementing one hour sepsis bundle assessed with checklist which were designed by four anesthsiologist-intensivists | upon study completion, in 1 day
  Measured by checklist which were designed by four anesthesiologist-intensivists before the study was conducted and validated by Aiken coefficient. The Aiken coefficient for this checklist were all >0.3 which is declared valid.

CONTACTS AND LOCATIONS:
Overall Officials: adhrie sugiarto, MD, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo General Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No